CLINICAL TRIAL: NCT01827605
Title: A Phase III Multicenter,Randomized Study Comparing Consolidation With 90yttrium-Labeled Ibritumomab Tiuxetan (Zevalin®) Radioimmunotherapy Vs Autologous Stem Cell Transplantation (ASCT) in Patients With Relapsed/Refractory Follicular Lymphoma (FL) Aged 18-65 Years
Brief Title: A Phase III Multicenter, Randomized Study Comparing RIT Vs ASCT in Patients With Relapsed/Refractory (FL)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_FLAZ-12
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Relapsed Follicular Lymphoma
Keywords: Relapsed follicular Lymphoma; RIT; Zevalin
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A RIT (Experimental): Infusion of 90Y Ibritumomab Tiuxetan if the patient has less than 25% BM infiltration at the pre-consolidation restaging (0.4 mCi/kg if platelets ≥150,000/mmc, 0.3 mCi/kg if platelets are between 100.000 and 150,000/mmc). Zevalin® will be delivered as per indications and should thus be provided at expenses following regular supplies procedures.
  Interventions: Other: ZEVALIN
- ARM B ASCT (Experimental): BEAM conditioning regimen (or in alternative FEAM regimen with fotemustine to replace BCNU) and reinfusion of CD34+ cells of ≥ 2x106/Kg CD34+ day 0 (optimal dose to reinfuse 4x106/Kg CD34+). G-CSF 5 mcg/Kg from day 2 until ANC>1500/mmc. Patients who failed mobilization will directly proceed to rituximab maintenance
  Interventions: Drug: BEAM

INTERVENTIONS:
Other: ZEVALIN — Infusion of 90Y Ibritumomab Tiuxetan if the patient has less than 25% BM infiltration at the pre-consolidation restaging (0.4 mCi/kg if platelets ≥150,000/mmc, 0.3 mCi/kg if platelets are between 100.000 and 150,000/mmc).
  Other Names: RIT
  Arms: Arm A RIT
Drug: BEAM — BEAM REGIMEN day -6 Carmustine* 300 mg/ m2 i.v. in 250ml dextrose 5% solution
  from day -5 to day -2 Cytarabine 200 mg/m2 i.v. every 12 hours in 250 ml dextrose 5% solution, 250 ml/hr Etoposide 100 mg/m2 i.v. every 12 hours in 250 ml dextrose 5% solution, 250 ml/hr day -1 Melphalan 140 mg/m2 i.v. in 100ml saline solution in 200 ml/hr
  day 0
  UReinfusion of autologous stem cells following this rules:
  1. Patient collecting ≥6x106 CD34+ cells/kg use >4x106 CD34+ cells/kg for ASCT and keep >2x106 CD34+ cells/kg for back up;
  2. Patient collecting 4-6x106 CD34+ cells/kg use >2x106 CD34+ cells/kg for ASCT and keep >2x106 CD34+ cells/kg for back up;
  3. Patient collecting 2-4x106 CD34+ cells/kg use all CD34+ cells for ASCT and keep no back up.
  day 2 Filgrastim or Lenograstim 5μg/Kg s.c. until ANC > 1500/mmc
  Other Names: ASCT
  Arms: ARM B ASCT

SUMMARY:
This is a Phase III, multicenter, open-label, randomized and controlled study to compare the efficacy of a consolidation therapy with RIT versus ASCT in patients with FL in CR or PR after second or third line chemotherapy supplemented with rituximab.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, open-label, randomized and controlled study to compare the efficacy of a consolidation therapy with RIT vs. ASCT in patients with FL in CR or PR after second or third line chemotherapy supplemented with rituximab. Patients with FL will be eligible for screening at the time of relapsed or refractory disease after two or less chemotherapy lines at least one containing rituximab.

This study will be conducted in six steps as follows. Screening Phase, Enrolment and Induction chemotherapy (STEP I) Randomization (STEP II) Stem cell mobilization and collection (STEP III) Consolidation (RIT vs ASCT) (STEP IV) Maintenance (STEP V) Follow-up Phase (STEP VI)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Histologically documented diagnosis of grade I-IIIa FL defined according to WHO guidelines 2008 (Re-biopsy required)
* Availability of BM and PB for Minimal Residual Disease (MRD) analysis (see Appendix I)
* Relapsed or refractory disease after ≤ two chemotherapy lines at least one containing Rituximab (Rituximab maintenance is UNOTU considered a therapeutic line)
* Clinical indication of treatment i.e. Stage II-IV who require therapy according to SIE and GELF criteria (see Appendix II)
* ECOG performance status 0-2 (unless disease-related) (see Appendix III)
* Availability of histological material for centralized revision
* Laboratory values:

  * ANC ≥ 1500/mmc unless due to marrow involvement by lymphoma and/or platelets ≥ 100000/mmc unless due to marrow involvement by lymphoma
  * Serum creatinine ≤ 1.5 x ULN, unless it is disease related
  * Bilirubin ≤ 1.5 x ULN (or ≤ 3.0 x ULN, if patient has Gilbert syndrome)
  * AST/SGOT and/or ALT/SGPT ≤ 2.5 x ULN if not lymphoma related or ≤ 5.0 x ULN in case of lymphoma liver involvement
* Adequate cardiac function: LVEF > 50% by echocardiography or MUGA scan
* Not pregnant or breast-feeding
* Willingness to use effective contraception during the study and 3 months after the end of treatment
* No other prior malignancies except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, or other cancer from which the patient has been disease-free for ≥ 5 years (see Exclusion criteria 14)
* Signed informed written consent

Exclusion Criteria:

* Grade IIIb FL, transformed FL or histologies different from FL
* Previous treatment with > two lines of chemotherapy ± rituximab Maintenance is UNOTU considered a therapeutics line)
* Previous ASCT or RIT treatment
* CNS involvement by lymphoma
* HBV positivity with the exception of patients who are seropositive because of hepatitis B virus vaccination and patients HbcAb positive and HbsAg negative with undetectable serum HBV-DNA. Occult carriers: must receive treatment with Lamivudine 100 mg for the duration of treatment program and at least 12 months after treatment cessation; HBV-DNA levels and HBsAg will be monitored every month
* HCV positivity with elevated transaminases or INR or APTT or active virus replication
* HIV positivity
* Any concurrent medical condition requiring long term use (> one month) of systemic corticosteroids
* Active bacterial, viral, or fungal infection requiring systemic therapy
* Any concurrent medical or psychiatric condition which might impair administration of therapy or preclude the ability to give informed consent
* Treatment with an experimental agent within 30 days prior to study entry
* Myelosuppressive chemo or biological therapy within three weeks before study entry (use rituximab course delivered as maintenance is not an exclusion therapy)
* Major surgery other than diagnosis within 4 weeks prior to study entry
* Previous i.v. or i.m. treatments with murine or animal derived antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-01; Primary Completion 2019-10 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival from randomization (rPFS) | 36 months
  PFS will be defined as the time between the date of randomization and the date of disease progression, relapse or death from any cause.

SECONDARY OUTCOMES:
Overall Survival from randomization (rOS) | 36 months
  OS will be defined as the time between the date of randomization and the date of death from any cause.
Event Free Survival (EFS) | 36 months
  EFS will be measured from the date of randomization to the date of any treatment failure including death, disease progression or relapse, discontinuation of treatment for any reason (toxicity, patient preference, initiation of new treatment without documented progression).
Treatment Free Survival from randomization (TFS) | 36 months
  TFS will be defined as the time between the date of the end of primary treatment until the institution of the next unplanned chemotherapy in randomized population.
Progression Free Survival from enrolment (ePFS) | 42 months
  PFS will be defined as the time between the date of enrolment and the date of disease progression, relapse or death from any cause.
Overall Survival from enrolment (eOS) | 42 months
  OS will be defined as the time between the date of enrolment and the date of death from any cause
Complete Response (CR) Rate | At the end of the consolidation phase (6 months)
  Proportion of CR according to the Cheson 2007 response criteria at the end of consolidation phase.
Overall Response Rate (ORR) | At the end of the consolidation phase (6 months)
  ORR at the end of the consolidation phase is defined as Complete Response (CR) or Partial Response according to the Cheson 2007 response criteria.
Toxicity | 42 months
  Incidence of grade 3 or higher Toxicity measured by CTCAE v.4.03 during therapy.
Molecular Response rate (MR) | 36 months
  Rate of MR will be defined as the proportion of patients achieving PCR negativity after the consolidation phase and during follow up.
Molecular Response rate conversion (cMR) | 6 months
  Rate of conversion will be defined as the proportion of patients with baseline PCR-positivity converting to PCR-negativity during treatment.
Molecular Relapse Rate (MRR) | 24 months
  Rate of molecular relapse will be defined as the proportion of patients with PCR-negativity after treatment converting to PCR-positivity during the first two years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, Principal Investigator — AO Città della salute e della Scienza di Torino - Ospedale S. Giovanni Battista - TORINO; Marco Ladetto, Principal Investigator — AO SS. Antonio e Biagio e Cesare Arrigo Alessandria
Locations (38):
- Italy (38):
  - A.O.U. San Martino, Genova, GE
  - Ematologia, A.O. San Gerardo, Monza, Milano
  - A.O. Niguarda, Milan, MI
  - IRCCS-Centro di riferimento oncologico UO di ematologia e Trapianto Cellule Staminali, Rionero in Vulture, Potenza
  - Azienda Ospedaliera "Bianchi Melacrino Morelli", Reggio Calabria, RC
  - Presidio Ospedaliero "A. Tortora", Pagani, SA
  - Emat Univ - Città della salute e della scienza di Torino, Torino, TO
  - Ospedale San Bortolo, Vicenza, VI
  - Ospedale Policlinico G.B. Rossi (Borgo Roma) Di Verona, Verona, VR
  - A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Clinica di ematologia AOU Umberto I Ospedali Riuniti, Ancona
  - Ematologia con Trapianto Policlinico Universitario Consorziale, Bari
  - Spedali Civili, Brescia
  - Presidio Ospedaliero A.Perrino - Divisione di Ematologia, Brindisi
  - Divisione di Ematologia Osp. Businco, Cagliari
  - IRCC Onco-Ematologia, Candiolo
  - Ospedale Ferrarotto, Catania
  - Policlinico Careggi Clinica Ematologica, Florence
  - A O Papardo, Messina
  - Ematologia e Trapianto IRCCS, Istituto Nazionale dei Tumori, Milan
  - IRCCS San Raffaele Unità di Chemioterapia, Milan
  - Policlinico di Modena - Università degli studi, Modena
  - Istituto Pascale Oncoematologia, Napoli
  - SCDU Ematologia - Università del Piemonte Orientale, Novara
  - Ospedale S. Francesco, Nuoro
  - Azienda Ospedaliera V. Cervello, Palermo
  - U.O. Complessa di Ematologia Ospedale di Parma, Parma
  - Ematologia Policlinico San Matteo, Pavia
  - Ospedale Santa Maria della Misericordia, Perugia
  - Ospedale Santo Spirito Dipartimento di Ematologia, Pescara
  - Unità Ematologia Ospedale Civile di Piacenza, Piacenza
  - Ausl Ravenna, Ravenna
  - SC Ematologia AO Santa Maria Nuova IRCCS, Reggio Emilia
  - Univeristà La Sapienza, Roma
  - SC Ematologia Città della salute e della scienza di Torino, Torino
  - Filippo Gherlizoni, Treviso
  - UO Ematologia Osp. Cardinale Panico, Tricase
  - Clinica di Ematologia - A.O.U. S. Maria di Udine, Udine